CLINICAL TRIAL: NCT06003335
Title: Increasing Physical Activity Through Personalised Motivational Messaging to Improve Cognitive Function in Lung Cancer Survivors With Cancer-related Cognitive Impairment: a Randomised Controlled Trial
Brief Title: Increasing Physical Activity Through Personalised Motivational Messaging to Improve Cognitive Function in Lung Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: uhongkongc9ttii37
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Neoplasms; Lung Cancer; Physical Inactivity; Cognitive Impairment
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Sedentary Behavior; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IG (Experimental): The intervention group will receive personalised motivational messages (according to their physical activity levels and preferences screened during the baseline measurement) using instant messaging applications (e.g., WhatsApp). They will be equipped with a wearable activity tracker for 3 months to monitor their physical activity level. In accordance with the guidelines for mobile instant messageing development, we will develop a message content library and protocol for intervention delivery.
  Interventions: Behavioral: Regular message delivery; Behavioral: Chat-type support message delivery
- CG 1 (Active Comparator): Control group 1 will receive regular message delivery (as mentioned in the intervention) without personalised motivational messaging for better evaluation of the effect of personalized motivational messaging.
  Interventions: Behavioral: Regular message delivery
- CG 2 (No Intervention): Control group 2 (self-management) will only receive a leaflet containing basic information about CRCI distributed during the recruitment process and text message reminders for follow-up surveys. Regular and real-time support (i.e., chat-type) messages will not be made available to the control group.

INTERVENTIONS:
Behavioral: Regular message delivery — Regular messages will be sent regularly to each participant over the 12-week study period. As personalisation is a core process in enabling behavioural change, the intervention content, frequency, and timing of the messages will be based on the participants' self-care needs and preferences, which will be surveyed at baseline. If no specific preferences are provided, we will plan the message delivery to decrease in frequency over time as this trend has shown the highest effectiveness in existing studies. The format of messages will be mainly texts, but other formats such as pictures and voice messages will also be considered for addition to the content library to suit a wide range of preferences.
  Arms: CG 1; IG
Behavioral: Chat-type support message delivery — Chat-based support will be given to the participants in addition to the regular message delivery. Instant messaging will be used to communicate directly with the participants. We plan to recruit 10 student RAs who have been trained in the delivery of interactive instant messages (IMs) to provide chat-type support to encourage increased physical activity and interaction. Participants will be invited to set physical activity goals and action plans through the chat-type support. Participants will receive a personalised summary of their physical activity weekly and will be encouraged to reflect on this through a real-time chat (around 5 minutes). They will also be encouraged to establish a plan of how they can adjust their physical activity goal going forward. When addressing the participants' queries or any ethical concerns, the student RAs will be instructed to immediately report to the Principal Applicant and supervisors who are experienced and trained research nurses.
  Arms: IG

SUMMARY:
Objectives: To examine the effectiveness of a personalised motivational messaging intervention for improving cognitive function in lung cancer survivors.

Hypothesis to be tested: Lung cancer survivors receiving personalised motivational messaging will have better cognitive function than usual care.

Design and subjects: A randomised controlled trial in 196 lung cancer survivors with cancer-related cognitive impairment.

Intervention: The intervention group will be equipped with a wearable activity tracker for 3 months and receive personalised motivational messages via instant messaging applications (e.g., WhatsApp) to promote physical exercise. The intervention will include 1) regular messages sent at preferred times and frequencies allowing participants to choose suggested physical activity goals, and 2) support via chat-type messaging such as goal setting, real-time counselling, and practical advice. The control group will receive a leaflet on cognitive impairment with reminder text messages for follow-up surveys.

Main outcome measures: Data will be conducted at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up). Primary outcome will be cognitive function measured by HK-MoCA (objective) and Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) scale (subjective). Secondary outcomes are physical activity (IPAQ-SF), self-efficacy for exercise (SEE), psychological well-being (PHQ-4), and quality of life (EORTC QLQ-C30).

Data analysis: Intention-to-treat, post-trial qualitative (compliance with the intervention), and cost-effectiveness analyses will be conducted. We will follow the CONSORT-EHEALTH checklist.

Expected results: This trial will provide evidence on the effectiveness of the proposed intervention on improving cognitive function and increasing physical activity among lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years;
2. diagnosed with stage I-III non-metastatic NSCLC cancer;
3. completed primary treatment with curative intent (surgery, chemotherapy and/or radiation therapy) 6 months to 5 years prior to the baseline assessment with no recurrence or occurrence of additional cancers;
4. identified as having mild cognitive impairment by the HK-MoCA 5-Min Protocol (≤ 7th age- and education-corrected percentile cut-off score);
5. not engaged in regular exercise (defined as < 150 min of moderate-intensity exercise per week).

Exclusion Criteria:

1. inadequate reading and verbal Cantonese comprehension for the study activities;
2. diagnosed with dementia;
3. unable to use mobile phone text messaging applications (e.g., WhatsApp).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Hong Kong Montreal Cognitive Assessment (HK-MoCA) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Primary outcome: objective cognitve function
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Primary outcome: subjective cognitve function

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Physical activity
Self-efficacy for exercise (SEE) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Self-efficacy for exercise
Patient Health Questionnaire 4 item (PHQ-4) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Psychological well-being
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | at baseline (T0), 3 months (T1; immediately after intervention delivery), and 6 months (T2; long-term follow up)
  Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho MH, Cheung DST, Tan JB, Lin CC. Ecological Momentary Mobile Cognitive Screening for Cancer-Related Cognitive Impairment Among Patients With Lung Cancer. Cancer Nurs. 2025 Jul 24. doi: 10.1097/NCC.0000000000001530. Online ahead of print. PMID 40711466